CLINICAL TRIAL: NCT00281190
Title: Innate and Adaptive Immunity in COPD Exacerbations: Clinically-Indicated Bronchoscopies
Brief Title: Comparison of Alveolar Macrophages in Individuals With COPD Versus Smokers With Normal Pulmonary Function
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey L. Curtis, Professor of Internal Medicine (Pulmonary & Critical Care Medicine), University of Michigan
Other Study IDs: 1326; R01HL082480 (NIH)
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy smokers: Smokers with normal pulmonary function
  Interventions: Procedure: Blood drawing; Procedure: Bronchoalveolar lavage during indicated bronchoscopy
- COPD patients: COPD patients
  Interventions: Procedure: Blood drawing; Procedure: Bronchoalveolar lavage during indicated bronchoscopy

INTERVENTIONS:
Procedure: Blood drawing — blood will be drawn at the time of starting the intravenous (IV) line for the procedure.
Procedure: Bronchoalveolar lavage during indicated bronchoscopy — A small amount of liquid will be introduced and immediately sucked back out of portions of the lung, and the cells that are recovered will be analyzed in the laboratory. All test will be solely for research, and there will be no results reported to the subject from that fluid.
  Other Names: BAL

SUMMARY:
The purpose of this study is to determine whether the alveolar macrophages (AMø) of patients with chronic obstructive pulmonary disease (COPD ) show abnormal responsiveness to bacterial and viral products, relative to smokers with normal pulmonary function. Participation in this study will be offered to patients already scheduled to undergo a bronchoscopy for clinical indications.

DETAILED DESCRIPTION:
BACKGROUND:

COPD is one of the most pressing healthcare problems facing our nation. Acute exacerbations of COPD (AE-COPD) are responsible for the bulk of healthcare costs, and much of the morbidity and decline in health status among individuals with this common disease. The lack of accepted animal models of AE-COPD necessitates novel approaches using human samples. Advances in the understanding of the pathogenesis have been slowed, in part, due to controversy as to how exacerbations should be defined. The prevailing paradigm has defined AE-COPD as event-based. Such definitions clearly identify groups of patients with accelerated loss of pulmonary function and increased mortality. However, limited data show that symptom-based definitions of AE-COPD also capture episodes inducing significant morbidity and functional decline, and hence of concern to patients. Fundamental mechanisms are lacking to explain AE-COPD defined by either means.

Controversy also surrounds triggers of AE-COPD. Bacteria and viruses are involved in some episodes, but the relative importance of each is intertwined with disputes over the definition of AE-COPD. Progress at linking specific pathogens to molecular pathogenesis has been slow, both due to their diversity, and to the high rates of bacterial colonization of patients with COPD, even in the stable state. Moreover, in many AE-COPD cases, no pathogen can be identified. Without negating the value of analyzing infections with specific species of pathogens, it appears that progress in molecular pathogenesis could be accelerated by focusing on unifying features of the pulmonary immune response during AE-COPD.

DESIGN NARRATIVE:

The purpose of this experiment is to determine whether the AMø of patients with COPD show abnormal responsiveness to bacterial and viral products, relative to smokers with normal pulmonary function. Specifically, the study will determine the dose-response characteristics of AMø from these two groups of subjects for production of interleukin (IL)-6, IL-18, and IL-23 (pro-inflammatory cytokines) on stimulation by purified Lipopolysaccharide, a synthetic lipopeptide (PAM3-Cys), or poly I:C. These stimuli mimic the response to Gram-negative bacteria, Gram-positive bacteria, and RNA viruses, respectively.

This research protocol involves adding a research bronchoalveolar lavage (BAL) to clinically indicated bronchoscopy that is being performed for evaluation of lung nodules suspected to possibly be malignant. The research BAL will be performed during the same procedure, but on the opposite lung from the radiographic lesion that motivated the bronchoscopy. Subjects will be COPD patients or smokers with normal pulmonary function recruited from the Pulmonary Clinic. Smoking history will be taken to mean at least 20 pack-years exposure, and could include current or ex-smokers. Bronchoscopy will be performed under conscious sedation using a fiberoptic bronchoscope, in almost all cases on outpatients (although stable inpatients could be considered for consent if they otherwise meet eligibility criteria). The setting is the Endoscopy suite at the Ann Arbor VA Hospital.

The procedures in this protocol involve the following upon enrollment: bronchoalveolar lavage (200 ml maximal instilled volume) and collection of blood for hematocrit, serum albumin, C-reactive protein, and IL-6.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of COPD and/or chronic bronchitis (study group, following American Thoracic Society guidelines)
* Willingness to participate in follow-up studies defined in the protocol
* Ability to give informed consent
* Already undergoing clinically indicated bronchoscopy

Exclusion criteria:

* Unstable cardiovascular disease
* Other systemic disease in which survival of more than 2 years is unlikely
* Mental incompetence or active psychiatric illness
* Currently taking more than 20 mg/day of Prednisone
* Participation in another experimental protocol within 6 weeks of study entry
* Asthma
* Cystic fibrosis
* Clinically significant bronchiectasis
* Lung cancer
* Other inflammatory or fibrotic lung disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Smokers with COPD or smokers with normal pulmonary function will be recruited from among subjects scheduled to undergo bronchoscopy for clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2005-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
alveolar macrophage functions in vitro | day of bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Curtis, Study Chair — University of Michigan at Ann Arbor
Locations (1):
- University of Michigan at Ann Arbor, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Freeman CM, Curtis JL, Chensue SW. CC chemokine receptor 5 and CXC chemokine receptor 6 expression by lung CD8+ cells correlates with chronic obstructive pulmonary disease severity. Am J Pathol. 2007 Sep;171(3):767-76. doi: 10.2353/ajpath.2007.061177. Epub 2007 Jul 19. PMID 17640964
- [Background] Freeman CM, Han MK, Martinez FJ, Murray S, Liu LX, Chensue SW, Polak TJ, Sonstein J, Todt JC, Ames TM, Arenberg DA, Meldrum CA, Getty C, McCloskey L, Curtis JL. Cytotoxic potential of lung CD8(+) T cells increases with chronic obstructive pulmonary disease severity and with in vitro stimulation by IL-18 or IL-15. J Immunol. 2010 Jun 1;184(11):6504-13. doi: 10.4049/jimmunol.1000006. Epub 2010 Apr 28. PMID 20427767
- [Background] Freeman CM, Martinez FJ, Han MK, Ames TM, Chensue SW, Todt JC, Arenberg DA, Meldrum CA, Getty C, McCloskey L, Curtis JL. Lung dendritic cell expression of maturation molecules increases with worsening chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Dec 15;180(12):1179-88. doi: 10.1164/rccm.200904-0552OC. Epub 2009 Sep 3. PMID 19729666
- [Background] Curtis JL, Todt JC, Hu B, Osterholzer JJ, Freeman CM. Tyro3 receptor tyrosine kinases in the heterogeneity of apoptotic cell uptake. Front Biosci (Landmark Ed). 2009 Jan 1;14(7):2631-46. doi: 10.2741/3401. PMID 19273223
- [Result] Punturieri A, Copper P, Polak T, Christensen PJ, Curtis JL. Conserved nontypeable Haemophilus influenzae-derived TLR2-binding lipopeptides synergize with IFN-beta to increase cytokine production by resident murine and human alveolar macrophages. J Immunol. 2006 Jul 1;177(1):673-80. doi: 10.4049/jimmunol.177.1.673. PMID 16785566
- [Result] Erb-Downward JR, Thompson DL, Han MK, Freeman CM, McCloskey L, Schmidt LA, Young VB, Toews GB, Curtis JL, Sundaram B, Martinez FJ, Huffnagle GB. Analysis of the lung microbiome in the "healthy" smoker and in COPD. PLoS One. 2011 Feb 22;6(2):e16384. doi: 10.1371/journal.pone.0016384. PMID 21364979
- [Result] Todt JC, Freeman CM, Brown JP, Sonstein J, Ames TM, McCubbrey AL, Martinez FJ, Chensue SW, Beck JM, Curtis JL. Smoking decreases the response of human lung macrophages to double-stranded RNA by reducing TLR3 expression. Respir Res. 2013 Mar 9;14(1):33. doi: 10.1186/1465-9921-14-33. PMID 23497334
- See also: COPD Foundation — http://www.copdfoundation.org/
- See also: Training Grant in Lung Diseases — http://www.med.umich.edu/intmed/pulmonary/edu/mtp.htm
- See also: Graduate Program in Immunology — http://www.med.umich.edu/immprog/